CLINICAL TRIAL: NCT02813083
Title: Detection of Pathological Lymphocytes in Patients With Autoimmune Disease
Status: Completed | Type: Observational
Sponsor: University of Minnesota (Other)
Responsible Party: Sponsor
Other Study IDs: 20494
Record Dates: First submitted 2016-06-22; First posted 2016-06-24 (Estimated); Last update posted 2024-04-05 (Actual); Status verified 2024-04

CONDITIONS: Arthritis, Rheumatoid
MeSH Terms: conditions — Arthritis, Rheumatoid

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Biospecimen Retention: Samples With DNA — Serum, peripheral blood mononuclear cells
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Rheumatoid Arthritis: Rheumatoid arthritis patients
  Interventions: Other: No intervention (observational)

INTERVENTIONS:
Other: No intervention (observational) — No intervention (observational)

SUMMARY:
This study will help the investigators design a method to detect the disease-causing immune cells in patients with rheumatoid arthritis (RA). Such methods are not currently available, but if successful, would help scientists to better understand the causes of RA.

DETAILED DESCRIPTION:
The investigators are interested in learning about the immune cells in the blood that contribute to disease in patients with rheumatoid arthritis (RA). They have developed a method for identifying a specific type of immune cells that can react against normal tissues in the body.

In this study, the investigators will enroll RA patients from the University of Minnesota clinics, collect blood samples from enrolled patients, and process the blood samples to isolate DNA, RNA, serum, and blood cells. They will use the serum to detect whether specific autoantibodies (Anti-cyclic Citrullinated Peptide, or anti-CCP) are present. In cases where anti-CCP antibodies are detected, the investigators may quantify the numbers of immune cells present that contain receptors with the same anti-CCP specificity. They may also test whether the numbers of immune cells with these receptors correlate with measures of disease activity in RA patients.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of rheumatoid arthritis

Exclusion Criteria:

* Use of rituximab immediately prior to visit
* Pregnancy

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The investigators will enroll 155 rheumatoid arthritis patients from the University of Minnesota Rheumatology clinics.
Sampling Method: Non-Probability Sample
Enrollment: 129 (Actual)
Dates: Start 2011-08 (Actual); Primary Completion 2023-09 (Actual); Study Completion 2023-09 (Actual)

PRIMARY OUTCOMES:
DAS28-ESR | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Mueller, M.D., Principal Investigator — University of Minnesota
Locations (1):
- University of Minnesota Department of Medicine, Minneapolis, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No